CLINICAL TRIAL: NCT01089101
Title: A Phase 1 and Phase II and Re-Treatment Study of AZD6244 for Recurrent or Refractory Pediatric Low Grade Glioma
Brief Title: Selumetinib in Treating Young Patients With Recurrent or Refractory Low Grade Glioma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03173; NCI-2012-03173 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PBTC-029B; CDR667932; PBTC-029 (Other: Pediatric Brain Tumor Consortium); PBTC-029 (Other: CTEP); U01CA081457 (NIH); UM1CA081457 (NIH); NCT01386450 (obsolete NCT alias)
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Low Grade Glioma; Recurrent Childhood Pilocytic Astrocytoma; Recurrent Neurofibromatosis Type 1; Recurrent Visual Pathway Glioma; Refractory Neurofibromatosis Type 1; Refractory Visual Pathway Glioma
MeSH Terms: conditions — Astrocytoma; Neurofibromatosis 1 | interventions — Specimen Handling; AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (selumetinib) (Experimental): Patients receive selumetinib PO BID on days 1-28. Cycles repeat every 28 days for up to 26 cycles in the absence of disease progression or unacceptable toxicity. Patients who experience a sustained objective response from selumetinib on the phase I or phase II portions of the trial, and who have completed 2 years of treatment and stopped study drug may be enrolled on the re-treatment study after progression/recurrence. Patients in the re-treatment study may continue treatment indefinitely in the absence of disease progression or unacceptable toxicities. Patients undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Selumetinib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Selumetinib — Given PO
  Other Names: ARRY-142886; AZD 6244; AZD-6244; AZD6244; MEK Inhibitor AZD6244

SUMMARY:
This phase I/II trial studies the side effects and the best dose of selumetinib and how well it works in treating or re-treating young patients with low grade glioma that has come back (recurrent) or does not respond to treatment (refractory). Selumetinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) or recommend a Phase II dose of AZD6244 (selumetinib) in children with recurrent or refractory low-grade glioma. (Phase I, completed as of April 29, 2013) II. To describe the toxicity profile and define the dose limiting toxicity of AZD6244 in children with recurrent or refractory low-grade glioma. (Phase I) III. To study the safety of the maximum tolerated dose (MTD) or recommended a Phase II dose (RP2D) of AZD6244 as determined based on safety data from children >= 12 years of age in children < 12 years of age; if the MTD/RP2D of the older children is too toxic for the younger children, we will de-escalate to one dose level below and study the safety of that dose in the younger age cohort. (Phase I) IV. To assess the sustained response rate of AZD6244 administered at 25 mg/m^2/dose twice daily (BID), in a single arm Phase II setting in patients assigned to strata based on neurofibromatosis (NF)-1 status and presence or absence of v-raf murine sarcoma viral oncogene homolog B (BRAF) aberrations, specifically BRAF V600E mutations and/or BRAF KIAA1549 fusion identified by immunohistochemistry (IHC) and fluorescence in situ hybridization (FISH), respectively. (Phase II, completed as of January 4, 2021) V. To estimate the sustained response rate and prolonged disease stabilization rate (defined as lack of disease progression for >= 12 courses) associated with AZD6244 in patients with recurrent and/or progressive low-grade gliomas who previously received treatment on PBTC-029 or PBTC-029B for a minimum of 12 courses, with at least stable disease or patients who had a sustained response but remained on treatment < 12 courses. (Re-treatment Study, enrollment complete as of April 23, 2019)

SECONDARY OBJECTIVES:

I. To characterize the inter- and intra-patient variability in AZD6244 pharmacokinetics administered on this schedule and to assess the influence of patient specific covariates (including concomitant drug therapy) on AZD6244 pharmacokinetics. (Phase I) II. To evaluate the feasibility of collecting pre-trial tumor samples and the feasibility of using in situ hybridization assay to identify BRAF aberrations in available tumor specimens. (Phase I) III. To determine if pre-trial tumor samples show the biochemical signature that indicates activation of the mitogen-activated protein kinase (MAPK) pathway. (Phase I) IV. To describe magnetic resonance imaging (MRI) characteristics of the tumors before and after treatment and to explore the diffusion changes in the tumors before and after treatment to determine if there is an early diffusion indicator of response. (Phase I) V. Within the constraints of a Phase I trial, to document antitumor activity of treatment with AZD6244, as measured by objective responses and progression-free survival (PFS). (Phase I) VI. To explore the pharmacogenetic polymorphisms in AZD6244 metabolizing enzymes and transporters and relate these polymorphisms to AZD6244 pharmacokinetics. (Phase I) VII. To estimate the PFS distributions associated with AZD6244 treatment separately in patients assigned to the six strata as well as for various other subsets e.g. histology and tumor grade across strata. (Phase II) VIII. To explore correlations between BRAF aberrations and treatment response and PFS in patients for whom relevant biology data are available. (Phase II) IX. To assess MAPK aberrations by a combination of whole-exome and ribonucleic acid (RNA) sequencing. (Phase II) X. To characterize the inter- and intra-patient variability in AZD6244 pharmacokinetics administered on this schedule at the MTD/RP2D. (Phase II) XI. To determine progression-free survival following re-treatment with AZD6244 for progressive, recurrent low-grade gliomas and to evaluate the impact of variables such as previous response, interval treatment regimens, BRAF status and previous dose of AZD6244. (Re-treatment Study) XII. To evaluate the toxicity profile of re-treatment with AZD6244 and correlate with toxicities seen during initial treatment. (Re-treatment Study) XIII. To evaluate the toxicity profile of re-treatment with AZD6244 beyond 2 years for those patients who continue to show benefit from the drug, i.e. at least stable disease (SD). (Re-treatment Study)

OUTLINE: This is a phase I dose-escalation study (completed as of April 29, 2013) followed by a phase II study.

Patients receive selumetinib orally (PO) twice daily (BID) on days 1-28. Cycles repeat every 28 days for up to 26 cycles in the absence of disease progression or unacceptable toxicity. Patients who experience a sustained objective response from selumetinib on the phase I or phase II portions of the trial, and who have completed 2 years of treatment and stopped study drug may be enrolled on the re-treatment study after progression/recurrence. Patients in the re-treatment study may continue treatment indefinitely in the absence of disease progression or unacceptable toxicities. Patient undergo blood sample collection on study.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Imaging evaluations necessary to establish eligibility for study entry must be done within three (3) weeks prior to registration
* All other evaluations necessary to establish eligibility for study entry must be done within two (2) weeks prior to registration
* Patients must start therapy within 7 calendar days of registration
* Laboratory values must be no older than seven (7) days prior to the start of therapy; if a test that is repeated after registration and prior to therapy is outside the limits for eligibility, it must be rechecked within 48 hours prior to the start of therapy; if laboratory values still fail to meet eligibility criteria, the patient may not receive protocol therapy
* All patients must meet the following inclusion and exclusion criteria; NO EXCEPTIONS WILL BE GIVEN
* Participant is willing to sign a screening consent and provide adequate pre-trial tumor material for BRAF testing (both for BRAF V^600E mutation and BRAF KIAA1549 fusion assessments)

  * All patients who are candidates for enrollment in stratum 5 based on their tumor histology must be pre-screened
  * Screening may be applied to potential stratum 1 and 2 patients
* Patients whose prior BRAF testing was performed at another lab (Clinical Laboratory Improvement Amendments [CLIA]/College of American Pathologist [CAP] certified or otherwise) must send additional tumor material to Brigham and Women's Hospital (BWH) for confirmation; however, to preserve available tumor material, patients whose tumor material has previously undergone BRAF analysis at the Lindeman and Ligon Labs at Brigham and Women's Hospital using the same procedures as described in this protocol, will not be required to submit additional tumor material for analysis; these patients must have both the BRAFV600E mutation and BRAF KIAA1549 fusion assessments done and if only one test was previously conducted; additional tissue will be required for the second test
* Patient must be >= 3 but =< 21 years of age at registration
* Patient must have one of the following:

  * For stratum 5: non NF-1 associated low grade glioma (LGG) (other than pilocytic astrocytoma or optic pathway glioma)
  * For stratum 1 or 2: non NF-1, non-optic pathway pilocytic astrocytoma; note: all patients with non NF-1 associated optic pathway glioma with or without tissue must be enrolled on stratum 4
* Patients with sporadic (non NF-1 associated), histologically diagnosed progressive, recurrent or refractory non-optic pathway pilocytic astrocytoma who have pre- treatment tumor tissue available for BRAF analysis
* NF-1 patients with radiographic evidence of a progressive, recurrent or refractory low grade glioma, with or without pre-treatment tumor tissue
* Patients with progressive, recurrent or refractory optic pathway glioma, with or without pre-treatment tumor tissue
* Patients with histologically diagnosed progressive, recurrent or refractory non NF-1 associated LGG (other than pilocytic astrocytoma or optic pathway glioma); these patients must have BRAF aberrations as documented by the Lindeman and Ligon Labs at Brigham and Women's Hospital using the same procedures
* Patients will be assigned to one of 6 strata prior to enrollment; all BRAF assessments used for stratification below must be done at the Lindeman and Ligon Labs at Brigham and Women's Hospital using the same procedures as described in this protocol; assessments for both BRAF V^600E mutation and BRAF KIAA1549 fusion are required for patients who will enroll on strata 1, 2 and 5

  * Stratum 1: patients with non NF-1 associated progressive, recurrent or refractory pilocytic astrocytoma with pre-trial tumor material available and with a BRAF aberration i.e. BRAFV^600E mutation and/or BRAF KIAA1549 fusion as determined by IHC and FISH, respectively; patients with optic pathway glioma are excluded
  * Stratum 2: patients with non NF-1 associated progressive, recurrent or refractory pilocytic astrocytoma with pre-trial tumor material available and without a BRAF aberration i.e. BRAF^V600E mutation and/or BRAF KIAA1549 fusion as determined by IHC and FISH, respectively; patients with optic pathway glioma are excluded
  * Stratum 3: patients with neuro-fibromatosis 1 (NF-1) associated progressive, recurrent or refractory low grade glioma (World Health Organization [WHO] grade I & II), with or without tissue
  * Stratum 4*: patients with non-NF1 associated progressive, recurrent or refractory optic pathway glioma with or without tissue available for BRAF evaluation
  * Stratum 5: patients with non NF-1 associated progressive, recurrent or refractory low grade glioma other than pilocytic astrocytoma or optic pathway glioma with a documented BRAF aberration identified in pre-trial tumor material
  * Stratum 6: patients with non-NF-1 associated progressive, recurrent or refractory low grade glioma (other than optic pathway glioma [OPG]) with tissue available for BRAF analyses who cannot be classified into stratum 1, 2 or 5 due to inadequate tissue quality, assay failure, etc

    * Clarification: Stratum 4 was specifically designed for patients with hypothalamic/optic pathway gliomas; the intent is that if there is any optic chiasm invasion regardless of where the tumor is originating from (chiasm vs. hypothalamus vs. other location), the patient should be enrolled on Stratum 4, regardless of whether the tumor has been biopsied or not; obviously, there are some tumors that include part of the hypothalamus and clearly do NOT include the chiasm at all; in these situations, and if the tumor is a biopsy proven pilocytic astrocytoma, these patients should be enrolled on Stratum 1 or 2 (depending upon BRAF status)
* Patients must have bi-dimensionally measurable disease defined as at least one lesion that can be accurately measured in at least two planes in order to be eligible for this study
* Patients must have received prior therapy other than surgery and must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, biologic therapy or radiotherapy prior to study entry
* Patients must have received their last dose of known myelosuppressive anticancer chemotherapy at least three weeks prior to study registration or at least six weeks if nitrosourea
* Patient must have received their last dose of the biologic agent >= 7 days prior to study registration

  * For biologic agents that have a prolonged half-life, at least three half-lives must have elapsed prior to registration
* Monoclonal antibody treatment: at least three half-lives must have elapsed prior to registration
* Radiation: patients must have:

  * Had their last fraction of local irradiation to primary tumor >= 12 months prior to registration; investigators are reminded to review potentially eligible cases to avoid confusion with pseudo-progression
  * Had their last fraction of craniospinal irradiation (> 24 Gy) > 3 months prior to registration
* Corticosteroids: patients who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to registration
* Patients must be off all colony-forming growth factor(s) for at least 1 week prior to registration (filgrastim, sargramostim, erythropoietin) and at least 2 weeks for long-acting formulations
* Patients must have a body surface area (BSA) >= 0.55 m^2
* Patients with neurological deficits should have deficits that are stable for a minimum of 1 week prior to registration
* Patients must be able to swallow capsules
* Karnofsky performance scale (KPS for > 16 years [yrs.] of age) or Lansky performance score (LPS for =< 16 years of age) >= 60 assessed within two weeks prior to registration
* Absolute neutrophil count >= 1,000/uL (unsupported) (within 14 days of registration and within 7 days of the start of treatment)
* Platelets >= 100,000/L (unsupported) (within 14 days of registration and within 7 days of the start of treatment)
* Hemoglobin >= 8 g/dL (may be supported) (within 14 days of registration and within 7 days of the start of treatment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal for age (within 14 days of registration and within 7 days of the start of treatment)
* Total bilirubin < 1.5 times upper limit of normal for age (within 14 days of registration and within 7 days of the start of treatment)
* Albumin >= 3 g/dL (within 14 days of registration and within 7 days of the start of treatment)
* Serum sodium and potassium within the institutional limits of normal (within 14 days of registration and within 7 days of the start of treatment)
* Serum calcium and magnesium above the institutional lower limit of normal (within 14 days of registration and within 7 days of the start of treatment)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73m^2 or a serum creatinine based on age as follows (within 14 days of registration and within 7 days of the start of treatment):

  * =< 5 years: 0.8 mg/dL
  * > 5 years but =< 10 years: 1 mg/dL
  * > 10 years but =< 15 years: 1.2 mg/dL
  * > 15 years: 1.5 mg/dL
* Left ventricular ejection fraction (LVEF) >= 55%
* Corrected QT (QTc) interval =< 450 msecs
* Hypertension:

  * Patients, 3-17 years of age must have a blood pressure that is =< 95th percentile for age, height and sex at the time of registration

    * The normal blood pressure by height, age and sex tables can be accessed in the Generic Forms section of the Pediatric Brain Tumor Consortium (PBTC) members' webpage
  * Patients who are >= 18 years of age must have a blood pressure that is < 140/90 mm of Hg at the time of registration
  * Note: if a blood pressure (BP) reading prior to registration is above the 95th percentile for age, height and sex it must be rechecked and documented to be =< the 95th percentile for age, height and sex prior to patient registration
* Female patients of childbearing potential must not be pregnant or breast-feeding; female patients of childbearing potential must have a negative serum or urine pregnancy test
* The effects of AZD6244 on the developing human fetus are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, and for four weeks after dosing with AZD6244 ceases; women of child-bearing potential must have a negative pregnancy test prior to entry; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; please note that the AZD6244 manufacturer recommends that adequate contraception for male patients should be used for 16 weeks post-last dose due to sperm life cycle
* Ability to understand and the willingness to sign a written informed consent document according to institutional guidelines
* ELIGIBILITY CRITERIA FOR ENROLLMENT ON THE RE-TREATMENT STUDY
* Patients must have recurrence or progression of their low-grade glioma after coming off treatment with AZD6244 on PBTC-029 or PBTC-029B, with or without having received additional anti-tumor therapy following discontinuation of AZD6244; the progression must be unequivocal and sufficient to warrant re-treatment in the opinion of the investigator; progression will be defined as either progressive disease (PD) that meets the study definitions of progressive disease by MRI or vision deterioration thought to be related to tumor in patients with optic pathway tumors
* Patients must have received treatment on PBTC-029 or PBTC-029B for a minimum of 12 courses with at least stable disease, or had a sustained response (partial response [PR]/ complete response [CR]) but remained on treatment < 12 courses
* Patients must have bi-dimensionally measurable disease defined as at least one lesion that can be accurately measured in at least two planes
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, biologic therapy or radiotherapy prior to study entry

  * Myelosuppressive chemotherapy: Patients must have received their last dose of known myelosuppressive anticancer chemotherapy at least three weeks prior to registration on the Re-treatment Study or at least six weeks if a nitrosourea
  * Biologic agent: Patient must have received their last dose of the biologic agent >= 7 days prior to study registration; for biologic agents and monoclonal antibody treatment, at least three half-lives must have elapsed prior to registration
  * Other investigational agents (not fitting into one of the above specified categories): patients must have received their last dose of any other investigational agent greater than 28 days prior to enrollment
  * Radiation: Patients must have:

    * Had their last fraction of local irradiation to the primary tumor >= 12 months prior to registration; investigators are reminded to review potentially eligible cases to avoid confusion with pseudo-progression;
    * Had their last fraction of craniospinal irradiation (> 24Gy) > 3 months prior to registration
  * Corticosteroids: Patients who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to registration
  * Growth factors: Patients must be off all colony-forming growth factor(s) for at least 1 week prior to registration (filgrastim, sargramostim, erythropoietin) and at least 2 weeks for long-acting formulations

Exclusion Criteria:

* Patients with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), likely interfere with the study procedures or results
* Patients taken off treatment for progressive disease on PBTC-029 or PBTC-029B
* Patients who are receiving any other anticancer or investigational agents
* Patients with uncontrolled seizures
* Previous mitogen-activated protein kinase (MEK) inhibitor use such as PD-0325901; CI1040; AS73026; GDC 0973; ARRY43182; GSK110212
* Prior treatment with a BRAF inhibitor such as vemurafenib or dabrafenib (previous treatment with sorafenib is allowed)
* Patients with other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome) that meets New York Heart Association (NYHA) class II or above
* Required use of a concomitant medication that can prolong the QT interval
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD6244
* Patients previously treated with a MEK inhibitor other than AZD6244

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 220 (Estimated)
Dates: Start 2010-07-07 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose and recommended phase 2 dose of selumetinib determined by dose-limiting toxicities (phase I) | 28 days
  Toxicities will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Stratum-specific objective response (complete response + partial response) rate sustained for 8 weeks (phase II) | 40 weeks
  For each stratum separately exact confidence interval estimates will be provided for the true, unknown rates of objective response. In addition, the confirmed sustained objective response rate observed during treatment by cumulative incidence functions will be estimated. This provides not only an overall estimate of the response rate but also an estimate of the timing of responses as a function of number of months of treatment.
Objective response (objective response = complete response + partial response) (re-treatment study) | Up to 48 weeks
  Exact confidence interval estimates will be provided.
Disease stabilization rates (re-treatment study) | At 1 year
  Disease stabilization rates will be measured.

SECONDARY OUTCOMES:
Plasma drug concentrations and pharmacokinetic parameters (Phase I) | Day 1 of cycle 1
  Plasma drug concentrations and pharmacokinetic parameters volume of the central compartment, elimination rate constant, half-life, apparent oral clearance, and area under the plasma concentration time curve.
Stratum-specific progression-free survival distribution (PFS) (phase II) | From the date of initial treatment to the earliest date of disease progression, second malignancy or death for subjects who fail; and to the date of last contact for subjects who remain at risk for failure assessed for up to 30 days
  Kaplan-Meier estimates of distributions of PFS all eligible subjects who received at least one dose of selumetinib will be provided separately for each stratum. It is unlikely that sufficient numbers of subjects will be followed until death to statistically support estimation of the survival distributions but survival estimation will also be considered.
Presence or absence of BRAF V600E mutations or BRAF KIAA1549 fusion (phase II) | Up to 30 days
  Will be assessed by immunohistochemistry and fluorescence in situ hybridization, respectively. Frequency tables summarizing the presence and absence of BRAF aberrations in all patients from whom tissue is available will be provided. The association of presence/absence and type of BRAF aberrations versus PFS will be explored via Kaplan-Meier-plots. Log-rank tests and/or Cox regression models may also be used to assess statistical associations between BRAF and PFS provided more than 10 events are observed in a given strata to make such assessments meaningful.
Progression-free survival (retreatment study) | From the date of re-treatment initiation to the earliest date of disease progression, second malignancy or death for patients who fail; and the last contact for patients who remain at risk for failure, assessed up to 30 days
  Kaplan-Meier estimates of progression-free survival distributions for all eligible patients will be provided. Exact confidence interval estimates will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Jason R Fangusaro, Principal Investigator — Pediatric Brain Tumor Consortium
Locations (17):
- United States (17):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Children's Memorial Outpatient Center in Lincoln Park, Chicago, Illinois
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Fangusaro J, Onar-Thomas A, Young Poussaint T, Wu S, Ligon AH, Lindeman N, Banerjee A, Packer RJ, Kilburn LB, Goldman S, Pollack IF, Qaddoumi I, Jakacki RI, Fisher PG, Dhall G, Baxter P, Kreissman SG, Stewart CF, Jones DTW, Pfister SM, Vezina G, Stern JS, Panigrahy A, Patay Z, Tamrazi B, Jones JY, Haque SS, Enterline DS, Cha S, Fisher MJ, Doyle LA, Smith M, Dunkel IJ, Fouladi M. Selumetinib in paediatric patients with BRAF-aberrant or neurofibromatosis type 1-associated recurrent, refractory, or progressive low-grade glioma: a multicentre, phase 2 trial. Lancet Oncol. 2019 Jul;20(7):1011-1022. doi: 10.1016/S1470-2045(19)30277-3. Epub 2019 May 28. PMID 31151904